CLINICAL TRIAL: NCT02637128
Title: In Vivo Efficacy of Artemether-Lumefantrine and Artesunate-Amodiaquine for Uncomplicated Plasmodium Falciparum Malaria in Malawi, 2014
Brief Title: In Vivo Efficacy of Artemether-Lumefantrine and Artesunate-Amodiaquine for Uncomplicated P. Falciparum Malaria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Kamuzu University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Malawi TES 2014
Record Dates: First submitted 2015-12-17; First posted 2015-12-22 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: MALARIA, FALCIPARUM
Keywords: MALARIA, FALCIPARUM; MALAWI; ARTEMETHER-LUMEFANTRINE; ARTESUNATE-AMODIAQUINE
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artemether, Lumefantrine Drug Combination; amodiaquine, artesunate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- artemether-lumefantrine (AL) (Experimental): 20mg artemether/120 mg lumefantrine per tablet, Coartem-D™; Novartis, Basel, Switzerland administered following manufacturer's prescribed weight-based dosing, twice daily for 3 days.
  5-14 kg: 1 tablet; 15-24: 2 tablets; 25-34 kg: 3 tablets; >34 kg: 4 tablets per dose
  Interventions: Drug: artemether-lumefantrine (AL)
- artesunate-amodiaquine (ASAQ) (Experimental): 25mg artesunate/67.5 mg amodiaquine or 50 mg artesunate/135mg amodiaquine per tablet, Coarsucam™; Sanofi-Aventis, Paris, France administered following manufacturer's prescribed weight-based dosing, once daily for 3 days 4.5-8.9 kg: 1 25mg/67.5 mg tablet; 9-17.9 kg: 1 50mg/135 mg tablet; 18-35.9 kg 2 50mg/135 tablets; >36 kg: 4 50mg/135mg tablets per dose
  Interventions: Drug: artesunate-amodiaquine (ASAQ)

INTERVENTIONS:
Drug: artemether-lumefantrine (AL) — Dispersible formulation of artemether-lumefantrine (Coartem-D™; 20mg artemether/120mg lumefantrine per tablet, Novartis, Switzerland) administered twice a day for 3 days according to manufacturer recommended dosing for weight
  Other Names: Coartem
  Arms: artemether-lumefantrine (AL)
Drug: artesunate-amodiaquine (ASAQ) — Co-formulated artesunate-amodiaquine (25mg artesunate/67.5mg amodiaquine and 50mg artesunate/135mg amodiaquine tablets) administered once a day for 3 days, according to manufacturer recommended dosing for weight
  Other Names: Coarsucam
  Arms: artesunate-amodiaquine (ASAQ)

SUMMARY:
This study was designed to determine the efficacy of both artemether-lumefantrine and artesunate-amodiaquine (but not to compare the efficacies of the two drugs) for the treatment of uncomplicated Plasmodium falciparum malaria at Machinga, Nkhotakota, and Karonga District Hospitals- Malawi.

DETAILED DESCRIPTION:
Background: Malaria is a cause of substantial morbidity and mortality in Malawi. Prompt and effective treatment of uncomplicated malaria remains a key strategy to reduce the public health burden of malaria. Due to the rising resistance to and declining efficacy of sulfadoxine-pyrimethamine, the first-line treatment for uncomplicated malaria from 1993 to 2007, the National Malaria Control Program (NMCP) revised the national treatment guidelines in 2007 and again in 2013. The revised treatment guidelines recommend artemether-lumefantrine as the first-line treatment for uncomplicated malaria and artesunate-amodiaquine as a second-line treatment for uncomplicated malaria. Data from Malawi suggests that these drugs remain efficacious. In a study conducted in 2004-2006 in Blantyre, artemether-lumefantrine was found to be efficacious. A more recent assessment of artemether-lumefantrine in vivo efficacy conducted in six sites in Malawi in 2009 also suggests that the standard formulation artemether-lumefantrine remains highly efficacious. In addition, both the dispersible formulation of artemether-lumefantrine (Coartem-D™) and artesunate-amodiaquine were extremely well tolerated and safe in studies conducted in Malawi as well as in other Sub-Saharan African countries. Given the potential for development of parasite resistance, it is imperative to continue to monitor the efficacy of these drugs as long as they remain the recommended treatment regimens.

Objective: Determine the efficacy of artemether-lumefantrine and co-formulated artesunate-amodiaquine for the treatment of uncomplicated Plasmodium falciparum malaria at Machinga, Nkhotakota, and Karonga District Hospitals- Malawi

Methods: A randomized drug efficacy trial will be conducted in Malawi. The trial will include 453 febrile children 6-59 months old with confirmed uncomplicated P. falciparum infection, seeking care at Machinga, Nkhotakota, and Karonga District Hospitals; 151 patients will be enrolled at each site (113 for artemether-lumefantrine and 38 for co-formulated artesunate-amodiaquine). Patients will be randomized to receive treatment with either the dispersible formulation of artemether-lumefantrine at a dose of 2/12 mg/kg body weight of artemether and lumefantrine, respectively, per dose, given twice a day for 3 days; or co-formulated artesunate-amodiaquine at a dose of 4 mg/kg/day artesunate and 10 mg/kg/day amodiaquine once a day for 3 days. Clinical and parasitological parameters will be monitored over a 28-day follow-up period to evaluate drug efficacy.

ELIGIBILITY:
Inclusion Criteria:

* age between 6 to 59 months
* mono-infection with P. falciparum detected by microscopy
* parasitaemia of 1,000-200,000/µl asexual forms
* presence of axillary temperature ≥ 37.5 °C or history of fever during the past 24 h
* ability to swallow oral medication
* ability and willingness to comply with the study protocol for the duration of the study and to comply with the study visit schedule
* informed consent from the parent or guardian of the child

Exclusion Criteria:

* presence of general danger signs in children aged 6-59 months or signs of severe falciparum malaria according to the definitions of World Health Organization
* mixed or mono-infection with another Plasmodium species detected by microscopy
* presence of severe malnutrition (defined as a child whose growth standard is below -3 z-score)
* presence of febrile conditions due to diseases other than malaria (e.g. measles, acute lower respiratory tract infection, severe diarrhoea with dehydration) or other known underlying chronic or severe diseases (e.g. cardiac, renal and hepatic diseases, HIV/AIDS)
* regular medication that may interfere with antimalarial pharmacokinetics
* history of hypersensitivity reactions or contraindications to any of the medicines being tested or used as alternative treatments

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 452 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Adequate clinical and parasitological response (ACPR) | 28 days
  Absence of parasitaemia on day 28, assessed by microscopy, irrespective of axillary temperature, in patients who did not previously meet any of the criteria of early treatment failure, late clinical failure or late parasitological failure

CONTACTS AND LOCATIONS:
Overall Officials: Don P Mathanga, MBBS, PhD, Principal Investigator — 1. Malaria Alert Centre (MAC), University of Malawi College of Medicine, Blantyre, Malawi
Locations (1):
- Malaria Alert Center, University of Malawi College of Medicine, Blantyre, Malawi, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: Undecided